CLINICAL TRIAL: NCT00697853
Title: Study to Evaluate the Immunogenicity and Safety of GSK Biologicals' Novel Adjuvanted Hepatitis B Vaccine Administered According to a 0, 6 Month Schedule and of Engerix™-B Administered According to a 0, 1, 6 Month Schedule in Healthy Adults
Brief Title: Immunogenicity and Safety of GSK Biologicals' HBV-MPL Vaccine (2 Doses), and of Engerix™-B (3 Doses) in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/030
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Adjuvanted hepatitis B vaccine; Recombinant hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

ARMS (5):
- Group A (Active Comparator)
  Interventions: Biological: Engerix™-B
- Group B (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group C (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group D (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group E (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129

INTERVENTIONS:
Biological: Engerix™-B — 3-dose intramuscular injection
  Arms: Group A
Biological: HBV-MPL vaccine 208129 — 2-dose intramuscular injection
  Arms: Group B; Group C; Group D; Group E

SUMMARY:
This study is undertaken to assess the immune response and safety profile of 4 lots of the novel adjuvanted hepatitis B vaccine that were formulated following different processes, with Engerix™-B as the control vaccine

DETAILED DESCRIPTION:
This is an open, randomized study with five groups, but the four groups receiving HBV-MPL candidate vaccine are double-blinded.

At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* A male or female between 15 and 50 years of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the subject and/or from the parents or guardians of the subject.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or use adequate contraceptive precautions for one month prior to vaccination and up to two months after the last vaccination

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine and ending 30 days after.
* Previous vaccination against hepatitis B.
* History of significant and persisting hematological, hepatic, renal, cardiac or respiratory disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrollment.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Oral temperature of ≥37.5°C (99.5°F).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration/ administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or intravenous drug abuse

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 1998-11; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At month 7

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | At months 1, 2 and 6
Occurrence and intensity of solicited local and general symptoms | 4-day follow-up period after each vaccination
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | 30-day follow-up period after each vaccination
Occurrence, intensity and relationship to vaccination of SAEs | Throughout the entire study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trial Call Center, Brussels, Belgium